CLINICAL TRIAL: NCT01814787
Title: Computer Automation for Diagnosis and Management of Childhood Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Aaron Carroll, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1R01DK092717 (NIH); 1R01DK092717 (NIH)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Pediatrics; Computerized Decision Support System
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHICA Type 2 Diabetes Module (Experimental): Children treated at the two intervention clinic sites will have be treated using the CHICA system AND will be provided access to the newly developed CHICA Type 2 Diabetes Module. The CHICA Type 2 Diabetes Module will assist pediatricians in identification of those children 10 years of age or older who are at increased risk for type 2 diabetes, it will provide pediatric physicians guidelines to screen for type 2 diabetes, and it will coordinate the diagnosis and long-term management of the condition.
  Interventions: Other: CHICA Type 2 Diabetes Module
- Usual Care (No Intervention): Those patients who are assigned to the control group will have the CHICA system but will NOT be cared for using the CHICA Type 2 Diabetes Module. The CHICA system will notify the physician of the child's BMI percentile on the physician worksheet. However, the CHICA system will not ask for any additional information related to risk factors for type 2 diabetes on the pre-screening form, no advice will be provided to the physician on the physician worksheet, nor will just-in-time documents or automated reminder calls be made available. Identification of patients at risk for type 2 diabetes and care of those patients will occur through routine practices for that clinic.

INTERVENTIONS:
Other: CHICA Type 2 Diabetes Module — Information with regard to family history of type 2 diabetes, race/ethnicity, and maternal history of gestational diabetes will be gathered for every patient. This data will then be utilized by the CHICA system when a child is age 10 or older and presents to the clinic. Data regarding the child's BMI at that time will be analyzed by the CHICA system. If the child's BMI > 85th percentile, a prompt will appear on the provider worksheet asking the clinician whether the child might have insulin resistance. All information will then be analyzed to determine whether the child has 2 or more risk factors for the development of type 2 diabetes. If at least 2 risk factors are present, then the CHICA system goes on to coordinate the diagnosis and long-term management of type 2 diabetes.
  Arms: CHICA Type 2 Diabetes Module

SUMMARY:
Increasing rates of type 2 diabetes among children and adolescents has considerable long-term implications not only for the affected individuals, but also for society and the health system as a whole. Pediatricians have unique and important opportunities to screen for type 2 diabetes and to promote lifestyle modification for those children identified with pre-diabetes; yet implementation of these practices within the pediatric primary care setting is far from ideal. The purpose of this study is to implement the ADA screening guidelines for type 2 diabetes and clinical management prompts within a pediatric primary care setting using a computer decision support system (CDSS) developed by the investigators research group - the Child Health Improvement through Computer Automation (CHICA) system. The investigators hypothesize that the coupling of CDSS with ADA guidelines will result in greater compliance with ADA recommended screening procedures as well as better clinical management of children identified as having pre-diabetes or type 2 diabetes.

DETAILED DESCRIPTION:
As the prevalence of obesity in the United States has risen, so too has the prevalence of type 2 diabetes, a disease typically associated with adults. The American Diabetes Association (ADA) has recommended screening children 10 years of age or older who are at substantial risk for the presence or development of type 2 diabetes. They also recommend that primary prevention efforts, such as lifestyle modification, be directed to high-risk children whose glucose levels are elevated but not yet diagnostic of diabetes. The choice of screening methodology remains controversial and implementation within the pediatric primary care setting is far from ideal. The purpose of this study is to implement the ADA screening guidelines for type 2 diabetes within pediatric primary care practices using a computer decision support system (CDSS) developed by the investigators research group - the Child Health Improvement through Computer Automation (CHICA) system. Using the CHICA system the investigators will also be implementing clinical management prompts for the pediatrician caring for children with risk factors for type 2 diabetes, with impaired fasting glucose (IFG), or with fasting glucose indicating the possibility of diabetes. One of the greatest strengths of the CHICA system is its ability to implement evidence-based recommendations from authoritative sources, in this case the ADA, in a format that integrates easily into routine pediatric care; the system can therefore overcome many of the barriers described by pediatricians to the screening of type 2 diabetes in children. While the use of CDSS is not new, its application within the pediatric population has not been as pervasive as in adult medicine. Moreover, the application of CDSS to the screening, diagnosis and management of type 2 diabetes in children is relatively unexplored. The specific aims for this study are to: (1) Expand and modify an existing computer-based decision support system (CHICA), to identify those children 10 years of age or older who are at increased risk for type 2 diabetes, to provide pediatric physicians guidelines to screen for type 2 diabetes, and to coordinate the diagnosis and long-term management of the condition and (2) Demonstrate both the feasibility and effectiveness of the CHICA Type 2 Diabetes Module to recognize those children in need of screening for type 2 diabetes and facilitate prompt diagnosis and management of the condition. Phase one (Aim 1) focuses on programming and enhancements to the CHICA system and will take 12 months to complete. Phase two consists of a randomized controlled trial conducted in four pediatric clinics in order to evaluate Aim 2. Randomization will be by clinic and the investigators hypothesize that the coupling of CDSS with ADA guidelines will result in greater compliance with ADA recommended screening procedures as well as better clinical management of children identified as having pre-diabetes or type 2 diabetes. Phase two will begin in year 2 and continue through quarter 2 of year 4. Phase three involves statistical analysis and manuscript preparation.

ELIGIBILITY:
Inclusion Criteria:

* A patient's chart will be eligible for chart abstraction if the child is age 10 or older and is a patient at one of the four clinics involved in the study.

Exclusion Criteria:

* None

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1369 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Carroll, MD, MS, Principal Investigator — Indiana University School of Medicine; Tamara Hannon, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hannon TS, Dugan TM, Saha CK, McKee SJ, Downs SM, Carroll AE. Effectiveness of Computer Automation for the Diagnosis and Management of Childhood Type 2 Diabetes: A Randomized Clinical Trial. JAMA Pediatr. 2017 Apr 1;171(4):327-334. doi: 10.1001/jamapediatrics.2016.4207. PMID 28192551

RESULTS

PARTICIPANT FLOW:
Groups:
- CHICA Type 2 Diabetes Module: Children treated at the two intervention clinic sites will have be treated using the CHICA system AND will be provided access to the newly developed CHICA Type 2 Diabetes Module. The CHICA Type 2 Diabetes Module will assist pediatricians in identification of those children 10 years of age or older who are at increased risk for type 2 diabetes, it will provide pediatric physicians guidelines to screen for type 2 diabetes, and it will coordinate the diagnosis and long-term management of the condition.
  CHICA Type 2 Diabetes Module: Information with regard to family history of type 2 diabetes, race/ethnicity, and maternal history of gestational diabetes will be gathered for every patient. This data will then be utilized by the CHICA system when a child is age 10 or older and presents to the clinic. Data regarding the child's BMI at that time will be analyzed by the CHICA system. If the child's BMI > 85th percentile, a prompt will appear on the provider worksheet asking the clinician
Period: Overall Study
Arm/Group | CHICA Type 2 Diabetes Module | Usual Care
Started | 685 | 684
Completed | 685 | 684
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CHICA Type 2 Diabetes Module: Children treated at the two intervention clinic sites will have be treated using the CHICA system AND will be provided access to the newly developed CHICA Type 2 Diabetes Module. The CHICA Type 2 Diabetes Module will assist pediatricians in identification of those children 10 years of age or older who are at increased risk for type 2 diabetes, it will provide pediatric physicians guidelines to screen for type 2 diabetes, and it will coordinate the diagnosis and long-term management of the condition.
  CHICA Type 2 Diabetes Module: Information with regard to family history of type 2 diabetes, race/ethnicity, and maternal history of gestational diabetes will be gathered for every patient. This data will then be utilized by the CHICA system when a child is age 10 or older and presents to the clinic. Data regarding the child's BMI at that time will be analyzed by the CHICA system.
- Total: Total of all reporting groups
Arm/Group | CHICA Type 2 Diabetes Module | Usual Care | Total
Number analyzed (Participants) | 685 | 684 | 1369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 685 | 684 | 1369
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344 | 313 | 657
  Male | 341 | 371 | 712
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 376 | 336 | 712
  Hispanic | 192 | 243 | 435
  White | 55 | 59 | 114
  Other/Unknown | 62 | 46 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Children With Documented Risk Factors for Type 2 Diabetes
Description: Number of children (ages 10 and older) with documented risk factors for type 2 diabetes (>85%BMI and 2 of 4 Risk Factors)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA Type 2 Diabetes Module | Usual Care
Number analyzed (Participants) | 685 | 684
Participants | 283 | 282

ADVERSE EVENTS:
Time Frame: two years
Description: Study progress and safety will be reviewed monthly. An annual report will be compiled and will include a list and summarization of adverse events. In addition, the annual report will address (1) whether adverse event rates are consistent with pre-study assumptions; (2) whether continuation of the study is justified on the basis that additional data are needed to accomplish the stated aims of the study; and (3) conditions whereby the study might be terminated prematurely.
Arm/Group | CHICA Type 2 Diabetes Module | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/685 | 0/684
Other Adverse Events (participants affected / at risk) | 0/685 | 0/684

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No